CLINICAL TRIAL: NCT03664700
Title: ADEPT 1 - Observational Study of the LMA Protector
Brief Title: Observational Study of the LMA Protector
Acronym: ADEPT1
Status: Terminated | Type: Observational
Why Stopped: Due to problems caused by the COVID-19 pandemic
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Royal United Hospital Bath NHS Trust (Other); Royal Berkshire NHS Foundation Trust (Other Government); Northampton General Hospital NHS Trust (Other); University Hospital of Wales (Other)
Responsible Party: Principal Investigator, Vassilis Athanassoglou, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 1338
Record Dates: First submitted 2018-07-26; First posted 2018-09-10 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Airway Complication of Anesthesia
Keywords: Supraglottic airway device; LMA Protector

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LMA Protector: The LMA Protector will be used
  Interventions: Device: LMA Protector

INTERVENTIONS:
Device: LMA Protector — The LMA Protector will be inserted when a supraglottic device is needed

SUMMARY:
The investigators want to investigate the user friendliness, and performance of the LMA Protector. The principal research question is to assess the overall performance of the LMA Protector. The investigators are merely making observations related to use of the device during clinical practice.

DETAILED DESCRIPTION:
There is a lack of research data on regarding the use of the LMA Protector. There is no regulatory requirement to collect or publish patient data on any device, either before CE marking or after. These devices are freely purchased and used.

There is, however, a professional duty to know that a device conforms to established norms for use. These norms are not official standards but rather, reference data against which a device can be clinically judged. Therefore, a device that is easy to insert but has a low 'leak pressure' (see above) is different from one that is more difficult to insert but as a high leak pressure. It is not that one is 'better' than the other, but rather that the data help create a 'usability profile' of the device which can be useful when making a clinical selection for the device.

Preoperative assessment:

During the preoperative visit, patient information leaflet will be given to the patients meeting the eligibility criteria.

Wherever possible, suitable patients will be identified in the preoperative assessment clinic and the information leaflet given. The patients will be given adequate time to read this information and any queries will be answered before being asked to sign a consent form. A detailed airway assessment will be performed by one of the investigators and documented on the study proforma.

Induction of anaesthesia:

On arrival in the anaesthetic room patients will be monitored with pulse oximetry, electrocardiography and invasive or non-invasive blood pressure measurements. After intravenous access is secured and the pre-surgical checklist completed, all patients will be pre-oxygenated using a facemask to achieve end tidal oxygen concentration of at least 80%. A 'sniffing' position of the head and neck and a 20 degree head-up bed tilt will be used for pre-oxygenation. General anaesthesia will be induced intravenously. After induction of anaesthesia, facemask ventilation will be commenced and anaesthesia maintained with an inhalational anaesthetic agent in oxygen or with total intravenous anaesthesia. The volatile agent's (anesthetic gases) concentration of 1 MAC adjusted for the patient's age will be achieved and maintained. This is normal process of anaesthesia applicable for all patients irrespective of participation in the study.

Supraglottic airway device (SAD) insertion:

Once deep plane of anaesthesia is confirmed, with the absence of movement to jaw thrust stimulation the SAD (LMA protector) will be inserted. The size of the device will be based on the manufacturer's recommendations for the body weight. The breathing system will be connected to the device. Ventilation of the lungs will be then confirmed by observing adequate bilateral chest inflation and square end-tidal capnogram wave with positive pressure ventilation. Adequate ventilation will be recorded if three tests are passed: 1) adequate chest movement, 2) an expired tidal volume of at least 7 ml/kg and 3) stable oxygenation. Time would continue until LMA® ProtectorTM inserted successfully. If it is not possible to insert the device or ventilate through it, two more attempts at placement of the device will be allowed. If placement has failed after two further attempts, the study will be abandoned and the other device will be used. If this fails on first attempt a different LMA or tracheal tube will be used as appropriate.

Maintenance of anaesthesia and recovery

The main interventions refer to the insertion of the airway device into the patient to obtain a airway and allow the conduct of the anaesthetic and therefore the surgery. However, if there are problems with the device and the airway obtained is suboptimal then the below interventions are allowed (which will be noted in the data collection form):

1. Neck extension - move patient's neck upward
2. Neck flexion - move patient's neck downward
3. Chin lift - manoeuvre to open the airway
4. Jaw thrust - manoeuvre to open the airway
5. Reposition of the device At the end of operation, anaesthetic agents will be discontinued while the device is left in place. The device will be removed after the patient has regained consciousness, and has responded to verbal command to open the mouth. Any complications that occur during the use of the device will be recorded.

Postoperative assessment Postoperatively in recovery or on the ward, the investigators will visit each patient and determine whether the following airway complications are present after surgery: sore throat (constant pain, independent of swallowing), dysphagia (difficulty in, or pain provoked by, swallowing), sore jaw, dysphonia (difficulty in, or pain on, speaking), numbness of the tongue or the oropharynx, ear pain, neck or mouth ache, hearing changes. Each complication will be graded as none, mild, moderate or severe. The same questions will be asked 24-48 hours later.

First visit During the first visit by the anaesthetist to the participant, at the anaesthetist's earliest opportunity, either in the recovery area or on the ward, the participants will be asked about the following complications, which will be graded as none, mild, moderate or severe.

1. Vomiting
2. Lip or tongue swelling
3. Hearing changes
4. Ear pain
5. Sore throat
6. Pain on swallowing
7. Jaw pain
8. Neck or mouth ache
9. Pain on speaking
10. Numbness of the tongue

Second visit (or telephone consultation) During the second visit 24-48 hours post-operatively on the ward or via telephone the participants will be asked about the following complications, which will be graded as none, mild, moderate or severe.

1. Vomiting
2. Lip or tongue swelling
3. Hearing changes
4. Ear pain
5. Sore throat
6. Pain on swallowing
7. Jaw pain
8. Neck or mouth ache
9. Pain on speaking
10. Numbness of the tongue

ELIGIBILITY:
Inclusion Criteria

* Adult participants who are having a general anaesthetic.
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* ASA 1 - 3 category patients
* Elective operations
* Urgent operations
* Patients suitable for an SAD based on patient and operation factors.

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

* Refusal of consent
* Age less than 18 years
* Require intubation for the operation
* Risk of regurgitation
* ASA 4 and above
* Mouth opening less than 2.5cm Require awake intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing operation under general anaesthesia with a supraglottic airway device
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Athanassoglou, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (5):
- United Kingdom (5):
  - Royal United Hospital, Bath
  - Aneurin Bevan University Health Board, Cardiff
  - Nothampton General Hospital, Northampton
  - Oxford University Hospitals, Oxford
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: No
Data will be collected prospectively on data collection sheets completed by the anaesthetist / investigator during anaesthesia. Each site will manage their own data set and the data will be pooled at the end of the recruitment phase across all sites. Data will be sent from sites to the lead study team only at the end of the data collection.
  Consent form and initial data collection forms will be filed in the master folder and kept locked in the dedicated research locker in the department. The PI at each site will have access to this log. Each site will assign a study ID for each participant and a record of these IDs will be kept in the site file. Only anonymised data will be sent from each trust to the main study team. No personal data will be sent to the coordinating centre.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LMA Protector
Started | 112
Completed | 111
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 50
  Ireland | 61

OUTCOME MEASURES:

1. Primary Outcome: First go Insertion Success Rate
Description: Whether insertion during first go was successful or not
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants | 100

2. Primary Outcome: First go Successful Ventilation Rate
Description: Whether ventilation during first go was successful or not
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants | 110

3. Primary Outcome: Number of Participants With Complication Free Insertions
Description: Number of participants with complication free insertions divided by total number of participants
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants | 72

4. Secondary Outcome: Time to First Square Capnography Waveform
Description: Record time in seconds of time to first capnography trace
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Seconds | 31 [26 to 40]

5. Secondary Outcome: Lowest Oxygen Saturation Level
Description: Record of lowest oxygen saturation reading across all participants
Time Frame: Day 1
Measure: Number; unit: Percent of oxygen saturation
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Percent of oxygen saturation | 91

6. Secondary Outcome: Interventions Needed to Ensure Airway Patency
Description: Collect number of predefined interventions needed to keep airway patent
Time Frame: Day 1
Population: The number analysed in one or more rows relates to the number of participants for whom 1 or more airway manipulations was required.
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants
  1 or more airway manipulation required | 67
  Manipulation: Jaw thrust: number analyzed (Participants) | 67
  Manipulation: Jaw thrust | 50
  Manipulation: Neck extension: number analyzed (Participants) | 67
  Manipulation: Neck extension | 45
  Manipulation: Chin lift: number analyzed (Participants) | 67
  Manipulation: Chin lift | 4
  Manipulation: Reposition device: number analyzed (Participants) | 67
  Manipulation: Reposition device | 3

7. Secondary Outcome: Number of Participants With Visible Chest Movement
Description: The success of ventilation will depend on whether there was visible chest movement
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants | 110

8. Secondary Outcome: Number of Participants With Adequate Tidal Volume at Attempt of Ventilation
Description: The success of ventilation will depend on whether there was tidal volume > 7ml/kg
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants | 110

9. Secondary Outcome: Number of Participants With Stable Oxygen Saturations
Description: The success of ventilation will depend on whether there was stable SpO2
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants | 110

10. Secondary Outcome: Number of Participants With Square Capnography Trace
Description: The success of ventilation will depend on whether there was square capnography trace
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants | 110

11. Secondary Outcome: Complications Occurrence During Insertion of Device, During Anaesthesia, and on Device Removal
Description: Collect number of pre-defined complications of device usage
Time Frame: Day 1
Population: Further breakdown of when complications occurred and the pre-defined complications of device usage are presented for the number of participants who experienced complications.
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants
  Number who experienced complications | 39
  Number who experienced complications immediately following device insertion: number analyzed (Participants) | 39
  Number who experienced complications immediately following device insertion | 6
  Number who experienced complications during maintenance of anaesthesia: number analyzed (Participants) | 39
  Number who experienced complications during maintenance of anaesthesia | 1
  Number who experienced complications upon extubation: number analyzed (Participants) | 39
  Number who experienced complications upon extubation | 32
  Number who experienced mucosal injury: number analyzed (Participants) | 39
  Number who experienced mucosal injury | 19
  Number who experienced mild post-operative sore throat: number analyzed (Participants) | 39
  Number who experienced mild post-operative sore throat | 37
  Number who experienced mild pain on swallowing: number analyzed (Participants) | 39
  Number who experienced mild pain on swallowing | 12
  Number who experienced mild post-operative dysphonia: number analyzed (Participants) | 39
  Number who experienced mild post-operative dysphonia | 7
  Number who experienced mild mouth pain: number analyzed (Participants) | 39
  Number who experienced mild mouth pain | 3
  Number who experienced mild jaw pain: number analyzed (Participants) | 39
  Number who experienced mild jaw pain | 3
  Number who experienced mild numbness of tongue: number analyzed (Participants) | 39
  Number who experienced mild numbness of tongue | 1

12. Secondary Outcome: Complications Occurrence During Insertion of Device, During Anaesthesia, and on Device Removal
Description: Collect number of pre-defined complications of device usage. Secondary complication where asked about on Day 2 to ensure patients had recovered from the effects of the anaesthetic and are able to report any complications.
Time Frame: Day 2
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | LMA Protector
Number analyzed (Participants) | 111
Participants
  Number who experienced complications | 13
  Vomiting: number analyzed (Participants) | 13
  Vomiting | 1
  Sore throat: number analyzed (Participants) | 13
  Sore throat | 10
  Pain on swallowing: number analyzed (Participants) | 13
  Pain on swallowing | 1
  Neck or mouth ache: number analyzed (Participants) | 13
  Neck or mouth ache | 1

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse events were collected upon removal of the device and upon questioning in the PACU.
Groups:
- LMA Protector: The LMA Protector will be used
  LMA Protector: The LMA Protector will be inserted when a supraglottic device is needed
  Major Complications (desaturation to 91%) 1; 0.9%
  Minor Complications 39, 35%
  * 6, 5.4% immediately following device insertion
  * 1, 0.9% during maintenance of anaesthesia
  * 32, 28.8% upon extubation
Arm/Group | LMA Protector
All-Cause Mortality (participants affected / at risk) | 0/111
Serious Adverse Events (participants affected / at risk) | 1/111
Other Adverse Events (participants affected / at risk) | 39/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMA Protector (N=111)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hiccoughing occurred immediately post induction followed by laryngospasm with desaturation to 91% for less than one minute.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMA Protector (N=111)
hiccoughing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Poor seal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Repositioning of device (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood on device (Respiratory, thoracic and mediastinal disorders) | 19 (19)
Pain on swallowing (Injury, poisoning and procedural complications) | 12 (12)
Tongue numbness (Injury, poisoning and procedural complications) | 1 (1)
Jaw pain (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03664700/Prot_SAP_000.pdf